CLINICAL TRIAL: NCT02026323
Title: Effect of Acupuncture on Insulin Sensitivity in Women With Polycystic Ovary Syndrome and Insulin Resistance: Study Protocol of a Prospective Observational Study
Brief Title: The Effect of Acupuncture on Insulin Sensitivity Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Yanhua-Zheng, Attending physician, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCOSAir
Record Dates: First submitted 2013-12-27; First posted 2014-01-01 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acupuncture (Experimental): "Normal weight" group,the PCOS women with insulin resistance who are normal weight( BMI=18.5-23Kg/m2).The acupuncture treatment will last for six months, 3 times per week, 30 minutes per treatment.
  Interventions: Other: acupuncture
- acupuncture 2 (Experimental): "Over weight or obese" group ,the PCOS women with insulin resistance who are overweight or obese: BMI >23 Kg/m2.The acupuncture treatment will last for six months, 3 times per week, 30 minutes per treatment.
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — acupuncture

SUMMARY:
Hyperinsulinemia and insulin resistance play a key role in the pathogenesis of polycystic ovary syndrome (PCOS). Insulin resistance is significantly associated with the long-term risks of metabolic syndrome and cardiovascular disease. Acupuncture with electrical stimulation has in rats with dihydrotestosterone (DHT)-induced PCOS been shown to improve insulin sensitivity. Whether these findings can be translated into women with PCOS has not been investigated. Therefore, this study aims to evaluate whether acupuncture improves insulin sensitivity, ovulation rate and quality of life in women with PCOS. Our hypothesis is that acupuncture with combined manual and low-frequency electrical stimulation of the needles improves insulin resistance, induces ovulation and improves quality of life.

DETAILED DESCRIPTION:
This is a prospective observational study. A total of 112 women with PCOS and insulin resistance will be recruited and randomized into two groups according to their body mass index (BMI), i.e. normal weight (BMI=18.5-23Kg/m2) group and overweight or obese (BMI > 23Kg/m2) group1. The acupuncture treatment will last for six months, 3 times per week, 30 minutes per treatment. The primary outcome is changes in insulin sensitivity from baseline to after 6 months of acupuncture treatment measured by OGTT.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. BMI ≥18.5Kg/m2
3. Confirmed diagnosis of PCOS according to the Rotterdam criteria: Oligo-, amenorrhea (less than 8 cycles per year) or/clinical or biochemical hyperandrogenism and/or polycystic ovarian morphology.
4. IR defined by the homeostatic model assessment (HOMA-IR: fasting insulin x fasting glucose/22.5) and 2.14 will be used as the cut off 33.
5. No desire of children and using barrier methods of contraception for 1 year.
6. Willing to sign the consent form

Exclusion Criteria:

1. With other endocrine disorders such as hyperprolactinemia (defined as two prolactin levels at least one week apart 25 ng/mL or greater or as determined by local normative values), nonclassic congenital adrenal hyperplasia (17-hydroxyprogesterone <3nmol/L), and androgen secreting tumors.
2. Patients with FSH levels > 15 mIU/mL. A normal level within the last year is adequate for entry.
3. Patients with uncorrected thyroid disease (defined as TSH < 0.2 mIU/mL or >5.5 mIU/mL). A normal level within the last year is adequate for entry.
4. Patients diagnosed with Type I diabetes, or Type I and Type II patients who receiving antidiabetic medications such as insulin, thiazolidinediones, acarbose, or sulfonylureas likely to confound the effects of study medication; patients currently receiving metformin for a diagnosis of Type I or Type II diabetes or for PCOS are also specifically excluded.
5. Patients with suspected Cushing's syndrome.
6. Use of hormonal or other medication including Chinese Herbal prescriptions which may affect the outcome at least in the past 3 months.
7. Pregnancy within the last 6 weeks.
8. Post-abortion or postpartum within last 6 weeks.
9. Breastfeeding within the last 6 months.
10. Patients received Acupuncture treatment related to PCOS within the last 2 months.
11. Patients who have undergone a bariatric surgery procedure in the recent past (<12 months) and are in a period of acute weight loss.
12. Patients with known congenital adrenal hyperplasia.
13. Not willing to give written consent to the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-10 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
HOMA-IR | baseline,treat for 3 and 6 month ,3 or 6 month follow-up

SECONDARY OUTCOMES:
FSH | baseline,up to 6 month,the follow-up of 3 or 6 month
  Determine FSH by electrogenerated chemiluminescence.
LH | baseline,up to 6 month,the follow-up of 3 or 6 month
Androgen | baseline,up to 6 month,the follow-up of 3 or 6 month
Progesterone | baseline,up to 6 month,the follow-up of 3 or 6 month
Prolactin | baseline,up to 6 month,the follow-up of 3 or 6 month
Estradiol | baseline,up to 6 month,the follow-up of 3 or 6 month
dehydroepiandrosterone(sodium)sulfate | baseline,up to 6 month,the follow-up of 3 or 6 month
sex hormone binding globulin | baseline,up to 6 month,the follow-up of 3 or 6 month
c-peptide | baseline,up to 6 month,the follow-up of 3 or 6 month
Apoa1 | baseline,up to 6 month,the follow-up of 3 or 6 month
ApoB | baseline,up to 6 month,the follow-up of 3 or 6 month
TC | baseline,up to 6 month,the follow-up of 3 or 6 month
TG | baseline,up to 6 month,the follow-up of 3 or 6 month
glycosylated hemoglobin | baseline,up to 6 month,the follow-up of 3 or 6 month
Questionnaire investigation | baseline,up to 6 month,the follow-up of 3 or 6 month
  Health related quality of life, affective symptoms and personality: Will be determined by short form-36 (SF36), polycystic ovary syndrome questionnaire (PCOSQ),(generic and diagnosis-specific HRQL questionnaire),and the Chinese Quality of Life (ChQOL) ,and symptoms of anxiety and depression assessed by the Zung Self-Rating Anxiety Scale (Zung SAS) and Zung Self-Rating Depression Scale (Zung SDS).
Transvaginal ultrasound | baseline,up to 6 month,the follow-up of 3 or 6 month

OTHER OUTCOMES:
Body composition(weight,height,waist circumference,hip circumference) | baseline,every month in treatment,the follow-up of 3 or 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia HX Ma, Dorctor, Study Chair — Study sponsor
Locations (1):
- The first affiliated hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Zheng YH, Wang XH, Lai MH, Yao H, Liu H, Ma HX. Effectiveness of abdominal acupuncture for patients with obesity-type polycystic ovary syndrome: a randomized controlled trial. J Altern Complement Med. 2013 Sep;19(9):740-5. doi: 10.1089/acm.2012.0429. Epub 2013 May 15. PMID 23676106
- [Derived] Zheng Y, Stener-Victorin E, Ng EH, Li J, Wu X, Ma H. How does acupuncture affect insulin sensitivity in women with polycystic ovary syndrome and insulin resistance? Study protocol of a prospective pilot study. BMJ Open. 2015 May 3;5(4):e007757. doi: 10.1136/bmjopen-2015-007757. PMID 25941189